CLINICAL TRIAL: NCT05009082
Title: Niraparib vs Niraparib in Combination With Bevacizumab in Patients With Carboplatinum-taxane Based Chemotherapy in Advanced Ovarian Cancer (A Multicentre Randomised Phase III Trial)
Brief Title: Niraparib vs Niraparib Plus Bevacizumab in Patients With Platinum/Taxane-based Chemotherapy in Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 28; 2024-516066-11-00 (EU CTIS Number); 2021-001271-16 (EudraCT Number); ENGOT-ov57 (Other: European Network for Gynecological Oncological Trial groups)
Record Dates: First submitted 2021-08-02; First posted 2021-08-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: High Grade Epithelial Ovarian Cancer; Advanced Ovarian Cancer; Niraparib; Bevacizumab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Chemotherapy followed by maintenance with niraparib
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Niraparib
- Arm 2 (Active Comparator): Chemotherapy in combination with bevacizumab followed by maintenance with bevacizumab and niraparib
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab; Drug: Niraparib

INTERVENTIONS:
Drug: Carboplatin — Area under curve (AUC) 5, intravenous, on day 1 every 3 weeks for 6 cycles
Drug: Paclitaxel — 175 mg/m², intravenous, on day 1 every 3 weeks for 6 cycles
Drug: Bevacizumab — 7.5 mg/kg or 15 mg/kg (according to local standard), intravenous, on day 1 every 3 weeks starting from cycle 2 in combination with chemotherapy and thereafter for up to 1 year starting from Cycle 7 Day 1
  Arms: Arm 2
Drug: Niraparib — 200 or 300 mg capsules once daily for up to a total of 3 years starting from Cycle 7 Day 1

SUMMARY:
This is an international, multicenter, randomized, open, Phase III trial to evaluate the efficacy and safety of carboplatin/paclitaxel/bevacizumab followed by bevacizumab and niraparib compared to carboplatin/paclitaxel followed by niraparib in patients with newly diagnosed advanced ovarian cancer.

DETAILED DESCRIPTION:
Eligible patients will be those patients with newly diagnosed, histologically confirmed, advanced (FIGO stage III/IV, except FIGO stage IIIA2 without nodal involvement) invasive high grade non-mucinous, non-clear cell epithelial ovarian cancer, peritoneal cancer, or fallopian tube cancer, who have either undergone upfront primary surgery or plan to undergo chemotherapy with interval debulking surgery (IDS). In addition, patients should not have any medical contraindications that would exclude treatment with bevacizumab and/or niraparib.

All eligible patients will receive the first cycle of chemotherapy (carboplatin area under curve [AUC] 5 and paclitaxel 175 mg/m²) as part of Study Run-In-Period (cycle 1). In parallel, central laboratory will determine the breast cancer (BRCA) status in tumor tissue (tBRCA). All patients with a valid central tBRCA test result will be randomized within 3 days prior to day 1 of cycle 2 in a 1:1 ratio in the following treatment arms:

Arm 1: Patients will receive further 5 cycles of carboplatin and paclitaxel q21d followed by niraparib once daily for up to a total of 3 years

Arm 2: Patients will receive further 5 cycles of carboplatin and paclitaxel plus bevacizumab q21d followed by bevacizumab q21d (for up to 1 year) and niraparib once daily for up to a total of 3 years.

The study aims to investigate, if the treatment strategy of carboplatin / paclitaxel / bevacizumab / niraparib is superior to the treatment of carboplatin / paclitaxel / niraparib-Inhibitor in an all-comer population.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the clinical trial requirements.
2. Female patients ≥ 18 years with histologically confirmed primary advanced invasive high grade non-mucinous, non-clear cell epithelial ovarian cancer, peritoneal cancer, or fallopian tube cancer FIGO III/IV (except FIGO stage IIIA2 without nodal involvement) according to recent FIGO classification (= FIGO stage IIIB - IV according to FIGO 2009 classification).
3. All patients must have had either upfront primary debulking surgery OR plan to undergo chemotherapy with interval debulking surgery.
4. Patients must have available tumor samples to be sent to central laboratory as formalin-fixed, paraffin-embedded (FFPE) sample for determination of BRCA status prior to randomization for stratification.
5. Patients must be able to commence systemic therapy within 8 weeks of cytoreductive surgery.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
7. Estimated life expectancy > 3 months.
8. Adequate bone marrow function (within 28 days prior to day 1, cycle 1 and within 3 days prior to day 1, cycle 2)

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L
   * Platelets (PLT) ≥ 100 x 10^9/L
   * Hemoglobin (Hb) ≥ 9 g/dL (can be post-transfusion)
9. Adequate coagulation parameters (within 28 days prior to day 1, cycle 1 and within 7 days prior to day 1, cycle 2)

   * Patients not receiving anticoagulant medication who have an International Normalized Ratio (INR) ≤ 1.5 and an Activated ProThrombin Time (aPTT) ≤ 1.5 x institutional upper limit of normal (ULN).
   * The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to institution medical standard) and the patient has been on a stable dose of anticoagulants for at least one week at the time of randomization.
10. Adequate liver and kidney function (within 28 days prior to day 1, cycle 1 and within 3 days prior to day 1, cycle 2)

    * Total bilirubin ≤ 1.5 x ULN (≤ 2.0 x ULN in patients with known Gilbert's syndrome) OR direct bilirubin ≤ 1.0 x ULN.
    * Aspartate aminotransferase / Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT) and Alanine aminotransferase / Serum Glutamic Pyruvate Transaminase (ALAT/SGPT) ≤ 2.5 x ULN, unless liver metastases are present, in case of liver metastases values must be ≤ 5 x ULN.
    * Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24 hour urine must demonstrate ≤ 1 g of protein in 24 hours.
    * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 30 mL/min (see Appendix 2).
11. Patients must have normal blood pressure (BP) or adequately treated and controlled BP, with a systolic BP of ≤ 140 mmHg and diastolic BP of ≤ 90 mmHg for eligibility. Patients must have a BP of ≤ 140/90 mmHg taken in the clinic setting by a medical professional within 4 weeks prior to day 1, cycle 1 and within 7 days prior to day 1, cycle 2.
12. Negative urine or serum pregnancy test within 7 days prior to day 1, cycle 1 in women of childbearing potential (WOCBP), confirmed prior to treatment on day 1.
13. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after administration of the last dose of medication.

    A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus).

    Examples of contraceptive methods with a failure rate of < 1% per year include but are not limited to bilateral tubal ligation and/or occlusion, male sterilization, and intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other clinical trial procedures, that include the completion of patient-reported outcomes questionnaires.

Exclusion Criteria:

1. Non-epithelial tumor origin of the ovary.
2. Ovarian tumors of low malignant potential (e.g. borderline tumors) and low grade tumors.
3. Planned intraperitoneal cytotoxic chemotherapy.
4. Malignancies other than ovarian cancer within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%) and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, ductal carcinoma in situ of the breast, or stage I p53 wild type endometrial cancer).
5. Prior systemic treatment for ovarian cancer.
6. Prior treatment with Poly adenosine diphosphate ribose polymerase (PARP) inhibitor.
7. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted).
8. Prior randomization in this trial.
9. Major surgery within 1 week of starting study treatment or patient who has not completely recovered from the effects of any major surgery. Core biopsy or other minor surgical procedure within 7 days prior to day 1, cycle 1 is permitted.
10. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to day 1, cycle 1) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to day 1, cycle 1) in case of suspected spinal cord compression.
11. Significant traumatic injury during 4 weeks preceding the potential first dose of bevacizumab.
12. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months prior to day 1, cycle 1.
13. History or evidence of thrombotic or hemorrhagic disorders within 3 months prior to day 1, cycle 1.
14. History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy e.g. uncontrolled seizures.
15. Pregnant or lactating women.
16. Treatment with any other investigational agent, or participation in another clinical trial testing a drug within 4 weeks or 5 times the half-life of the drug, whichever is longer, prior to day 1, cycle 1 or concomitantly within this trial.
17. Known hypersensitivity to bevacizumab and its excipients, Chinese hamster ovary cell products or other recombinant human or humanized antibodies. Known hypersensitivity to niraparib, paclitaxel and carboplatin and its components or excipients.
18. Non-healing wound, active ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no severe evidence of facial dehiscence or infection are eligible; regular wound examination will be performed.
19. Clinically significant cardiovascular disease, including

    * Myocardial infarction or unstable angina within 6 months of day 1, cycle 1
    * New York Heart Association (NYHA) Grade 2 Congestive Heart Failure (CHF),
    * Poorly controlled cardiac arrhythmia despite medication (patients with rate-controlled atrial fibrillation are eligible)
    * Grade ≥ 3 peripheral vascular disease (i.e. symptomatic and interfering with activity of daily living (ADL) requiring repair or revision)
    * Significant vascular disease including aortic aneurysm requiring surgical repair
20. Pre-existing sensory or motor neuropathy ≥ Grade 2.
21. (Intentionally left blank)
22. Patients with a history of or current Nephrotic syndrome.
23. Persistent cancer-related bowel obstruction (including subocclusive disease). Patients with a known history of ileus, who have been successfully treated and who are free of symptoms, may be eligible after consultation of sponsor.
24. History of abdominal fistula or tracheoesophageal fistula or gastrointestinal perforation or active gastrointestinal bleeding or anastomotic insufficiency within 6 months of day 1, cycle 1.
25. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of niraparib.
26. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
27. Any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
28. Previous allogeneic bone marrow transplant or previous solid organ transplantation.
29. Current or recent (within 10 days prior to day 1, cycle 1) chronic use of aspirin > 325 mg/day. Patients treated with other inhibitors of platelet aggregation such as clopidogrel, prasugrel, ticlopidine, tirofibane or dipyridamole should not be included into the trial.
30. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. This includes also any psychiatric disorder that prohibits obtaining informed consent.
31. Patient has known active hepatitis B or hepatitis C.
32. Patient has a history of Posterior Reversible Encephalopathy Syndrome (PRES).
33. Patients with chronic inflammatory bowel disease and active treatment for disease control.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Assessed frequently during the trial until observation of 586 PFS events or three years after Last Patient In, whichever occurs earlier
  Defined as the time from randomization to first progressive disease (PD) or death, whichever occurs earlier. PD is based on investigators assessment using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

SECONDARY OUTCOMES:
PFS according to tumor BRCA status | Assessed frequently during the trial until observation of 586 PFS events or three years after Last Patient In, whichever occurs earlier
  Defined as the time from randomization to first progressive disease (PD) or death, whichever occurs earlier. PD is based on investigators assessment using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Overall Survival (OS) | at every visit during the trial up to 66 months after Last Patient In
  Defined as the time from randomization to death
Time to First Subsequent Therapy (TFST) | at every visit during the trial up to 66 months after Last Patient In
  Defined as the time from randomization to the first subsequent treatment or death, whichever occurs earlier
Second Progression (PFS 2) | at every visit during the trial up to 66 months after Last Patient In
  Defined as the time from randomization to the second progression or death, whichever occurs earlier
Time to Second Subsequent Therapy (TSST) | at every visit during the trial up to 66 months after Last Patient In
  Defined as the time from randomization to the second subsequent treatment death whichever occurs earlier
Number of participants with treatment-related adverse events (AE) and/or serious adverse events (SAEs) and/or AEs that led to premature withdrawal of trial treatment and/or interruptions/dose modifications | at every visit during the trial up to safety follow up visit 30 days after last dose
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Effects on Quality of Life (QoL) | Assessed frequently during the trial up to 66 months after Last Patient In
  Questionnaires to be completed by patients and collected frequently during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, MD, PhD, Study Chair — KEM Essen | Evang. Kliniken Essen-Mitte gGmbH
Locations (65):
- Germany (65):
  - Klinikum St. Marien Amberg, Amberg
  - Klinikum Augsburg, Augsburg
  - Hochtaunus-Kliniken, Bad Homburg
  - Helios Klinikum Berlin-Buch, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Städt. Klinikum Brandenburg, Brandenburg
  - Klinikum Bremen Mitte, Bremen
  - Klinikum Chemnitz, Chemnitz
  - St. Elisabeth-Krankenhaus Köln-Hohenlind, Cologne
  - Klinikum Dortmund, Dortmund
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Florence-Nightingale-Krankenhaus Düsseldorf, Düsseldorf
  - Universitätsfrauenklinik Düsseldorf, Düsseldorf
  - KEM Essen | Evang. Kliniken Essen-Mitte gGmbH, Essen
  - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt am Main
  - Universitätsklinikum Gießen, Giessen
  - Klinikum Gütersloh, Gütersloh
  - Universitätsklinikum Halle, Halle
  - Albertinen Krankenhaus, Hamburg
  - Mammazentrum HH am Krankenhaus Jerusalem, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Gynäkologisch-Onkologische Praxis am Pelikanplatz, Hanover
  - Universitätsklnikum Heidelberg, Heidelberg
  - Klinikum am Gesundbrunnen / SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Gyn.-onkolog. Gemeinschaftspraxis Hildesheim, Hildesheim
  - Universtitätsklinikum Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - Klinikverbund Kempten-Oberallgäu gGmbH, Kempten
  - Klinikum Konstanz, Konstanz
  - Zentrum für ambulante gynäkologische Onkologie am HELIOS Klinikum Krefeld, Krefeld
  - Universitätsklinikum Leipzig, Leipzig
  - St. Vincenz Krankenhaus, Limburg
  - Klinikum Ludwigsburg, Ludwigsburg
  - UKSH Campus Lübeck, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - UKGM Gießen/Marburg Standort Marburg, Marburg
  - Mühlenkreiskliniken, Johannes Wesling Klinikum Minden, Minden
  - LMU Klinikum München-Großhadern, München
  - Rotkreuzklinikum München, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Neumarkt, Neumarkt
  - MVZ Nordhausen, Nordhausen
  - Ortenau Klinikum Offenburg-Kehl, Offenburg
  - St. Vincenz Krankenhaus GmbH, Paderborn
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Klinikum am Steinenberg, Reutlingen
  - RoMed Klinikum Rosenheim, Rosenheim
  - Klinikum Südstadt Rostock, Rostock
  - Thüringen-Kliniken "Georgius Agricola", Saalfeld
  - Leopoldina Krankenhaus Schweinfurt, Schweinfurt
  - g.SUND, Stralsund
  - Klinikum Stuttgart, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Klinikum Mutterhaus, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinik Ulm, Ulm
  - St. Josefs-Hospital, Wiesbaden
  - Klinikum Worms, Worms

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heitz F, Marth C, Henry S, Reuss A, Cibula D, Gaba Garcia L, Colombo N, Schmalfeld B, de Gregorio N, Wimberger P, Hasenburg A, Sehouli J, Gropp-Meier M, Schouten PC, Hahnen E, Hauke J, Polleis S, Harter P. AGO-OVAR 28/ENGOT-ov57. Niraparib alone versus niraparib in combination with bevacizumab in patients with carboplatin-taxane-based chemotherapy in advanced ovarian cancer: a multicenter randomized phase III trial. Int J Gynecol Cancer. 2023 Dec 4;33(12):1966-1969. doi: 10.1136/ijgc-2023-004944. PMID 37935524
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961